CLINICAL TRIAL: NCT03867786
Title: The Acute Effects of Resistance Exercise on Cannabis Use and Craving
Brief Title: Resistance Exercise and Cannabis Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Gwendolyn Thomas, Assistant Research Professor, Kinesiology, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2018-02-11; First posted 2019-03-08 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cannabis Use Disorder
Keywords: Resistance Exercise Neurobiological Mechanisms
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Condition (Experimental): Participants will undergo a 40 minute exercise protocol
  Interventions: Behavioral: Exercise
- Video Control Condition (Active Comparator): Participants will view a 40 minute nature video
  Interventions: Behavioral: Video Control

INTERVENTIONS:
Behavioral: Exercise — Participants will complete an acute exercise visit.
  Arms: Exercise Condition
Behavioral: Video Control — Participants will complete a video control visit.
  Arms: Video Control Condition

SUMMARY:
Cannabis is the most widely used illicit drug and rates of hazardous use, and cannabis use disorders (CUDs), have continued to rise in recent years. The highest rates of use and CUDs are seen in young adults (20 - 24 years old) with more than 50% of young adults reporting lifetime use of cannabis, 35% report use in the past year, and 20% report use in the past month. Increased exposure produces higher risk for detrimental psychological and behavioral effects of cannabis use. Given this increased prevalence of cannabis use and associated risks, identifying effective behavioral strategies that reduce cannabis craving, negative psychological effects, and alter neurobiological mechanisms underlying problematic cannabis use are an avenue of needed research. Exercise, particularly resistance exercise, is a behavioral intervention with considerable potential as an adjunctive treatment for CUD.

DETAILED DESCRIPTION:
Cannabis is the most widely used illicit drug and rates of hazardous use, and cannabis use disorders (CUDs), have continued to rise in recent years. The highest rates of use and CUDs are seen in young adults (20 - 24 years old) with more than 50% of young adults reporting lifetime use of cannabis, 35% report use in the past year, and 20% report use in the past month. Increased exposure produces higher risk for detrimental psychological and behavioral effects of cannabis use. Given this increased prevalence of cannabis use and associated risks, identifying effective behavioral strategies that reduce cannabis craving, negative psychological effects, and alter neurobiological mechanisms underlying problematic cannabis use are an avenue of needed research. Exercise, particularly resistance exercise, is a behavioral intervention with considerable potential as an adjunctive treatment for CUD.

The aims of this proposal seek to address these issues by implementing acute resistance exercise protocol in men and women who have cannabis use disorder. This proposal will: 1 examine the effect of an acute resistance exercise protocol on affect, stress, and compulsive urge to use in non-treatment seeking young adults with CUD 2.examine whether an acute resistance exercise session in individuals with CUD is associated with induced alterations in the appetitive/ reward hormone ghrelin These findings will inform the further development for exercise interventions for cannabis use disorder that can be used with the aim of supporting individuals with CUD reduce use and decrease the negative effects of withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals between the ages of 18-30 years who currently meet for a moderate or severe cannabis use disorder according to DSM-5 criteria.
2. Untrained (no structured exercise program for at least the previous 6 months) as verified by self-report on a physical activity form.
3. No previous bone or muscle problems or previous injuries that would prevent free movement about the shoulder, hip, knee or ankle, or increase the risk of discomfort or injury during exercise. No ongoing back problems.
4. No known endocrine disorders (including, but not limited to Hyperthyroidism, Hypothyroidism, Hyperparathyroidism, Cushing's Syndrome, Diabetes mellitus, metabolic syndrome or other inflammatory disorders).
5. No history of blood clotting disorders.
6. Able to read English and complete study assessments
7. Voluntarily provide informed consent and sign the informed consent document.
8. Able to provide negative toxicology screenings for substances, except for cannabis, at intake.

Exclusion Criteria:

1. Meet current criteria for a moderate or severe substance use disorder for any other substance besides cannabis
2. Have any current psychiatric disorders with acute symptoms (i.e., psychosis, suicidal, homicidal, current mania).
3. Younger or older than the specified age range of 18-30.
4. Any endocrine, bone, muscle problems, previous injuries, back problems, or blood clotting disorders.
5. Cardiac and severe respiratory illnesses (i.e. arrhythmias, enlarged heart, COPD) -

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Cannabis Craving | change from baseline
  Craving Marijuana Craving Questionnaire (MCQ) The 45-item MCQ is a multi-dimensional questionnaire that assesses marijuana craving. It is based on the the Cocaine Craving Questionnaire and uses items that touch on four specific constructs characterizing craving for marijuana: (1) compulsivity, an inability to control marijuana use; (2) emotionality, use of marijuana in anticipation of relief from withdrawal or negative mood; (3) expectancy, anticipation of positive outcomes from smoking marijuana; and (4) purposefulness, intention and planning to use marijuana for positive outcomes. Each item is rated on a seven-point Likert-type scale ranging from "strongly agree to strongly disagree"
Cannabis Craving | Change from baseline
  Total Ghrelin as measured by 0.5mL plasma
Cannibis Consumption | change from Baseline
  endocannabinoid N-arachidonoylethanolamine (AEA)

IPD SHARING:
Plan to Share IPD: Undecided